CLINICAL TRIAL: NCT04199806
Title: Retrospective Study of Patient Surveys of MMS Experience
Brief Title: Retrospective Study of Patient Surveys
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This is a retrospective study reviewing subject questionnaires. No treatments will be administered in this study.
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA19-004
Record Dates: First submitted 2019-12-03; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Questionnaire Review (Other)
  Interventions: Other: Questionnaire review

INTERVENTIONS:
Other: Questionnaire review — Review data from questionnaires received about MMS experience.

SUMMARY:
To collect data from Allergan Patient Surveys (patient surveys) and Allergan Patient Information Form (patient information form) to describe:

1. Patient demographics
2. Treatment patterns
3. Patient feedback and overall experience with MMS treatment

ELIGIBILITY:
Inclusion Criteria

* Subject has received MMS treatment in the abdomen and/or buttocks (with CoolTone prototype)
* Subject has completed the Allergan patient survey and information form on MMS experience between July 1, 2019 and December 1, 2019.

Exclusion Criteria

• There are no exclusion criteria for this study.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy Endpoint: Overall Experience Questionnaire | Immediately post subjects final treatment.
  Evaluation of patient overall experience with MMS treatment as measured by patient survey.

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie Jiang, NP, Study Director — Zeltiq Aesthetics

IPD SHARING:
Plan to Share IPD: No